CLINICAL TRIAL: NCT00768313
Title: A Multi-Centre Randomized Phase IV Clinical Trial Comparing Rods of Varying Yield Strengths and Their Ability to Hold Correction of Adolescent Idiopathic Scoliosis.
Brief Title: Phase IV Comparing Rods of Yield Strengths to Correct Adolescent Idiopathic Scoliosis.
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: Queen's University (Other)
Collaborators: DePuy Orthopaedics (Industry)
Responsible Party: Principal Investigator, Dr. Daniel Borschneck, Principal Investigator, Queen's University
Allocation: Randomized | Masking: Single | Purpose: Other
Other Study IDs: DB-012008
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Scoliosis
Keywords: scoliosis correction rod strength adolescent
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: titanium rod — comparison of rods of varying yield strengths and their ability to hold correction of scoliosis.
Device: ultra strength stainless steel rod — interventions involving rods of various strength to treat scoliosis
  Other Names: Expedium ultra strength stainless steel rod (220KSI).

SUMMARY:
There has been a growing trend amongst surgeons to use a construct for correction of scoliosis which involves segmental instrumentation with pedicle screws. Pedicle screw proponents cite greater curve control in all planes, which results in improved spinal curve correction. Some surgeons have noted due to the increased strength of the all screw construction that the rod is now the weak part of the spinal fixation. Although no evidence has been raised in regards to hardware failure there is a perception that a loss of balance in the sagittal plane is the result of flex in the titanium rod. A novel solution to the issue of rod flexibility is raised with the expedium super steel instrumentation which allows for greater stiffness than a 5.5 mm titanium rod with the same lower profile. This study aims to compare the new super steel technology with other established instrumentations used to correct spinal stenosis.

DETAILED DESCRIPTION:
screw purchase was to be recorded but study has been withdrawn.

ELIGIBILITY:
Inclusion Criteria:

* aged 10-20;
* presenting with a progressive lenke type 1A, N; or
* type idiopathic adolescent scoliosis measuring greater than 45 degree cobb angle

Exclusion Criteria:

* rigid scoliosis requiring a three column release or osteotomy;
* patients that can not have pedicle screw instrumentation due to technical concerns

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
percent correction in both frontal and sagittal planes for idiopathic scoliosis | pre-op, 3, 6, 12, 24 months

SECONDARY OUTCOMES:
screw purchase | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Borschneck, MD, Principal Investigator — Queen's Univeristy
Locations (1):
- Queen's Univeristy, Kingston, Ontario, Canada